CLINICAL TRIAL: NCT05323123
Title: Preparing for Pre-exposure Prophylaxis Implementation in Central-Eastern European Countries With Low Access to Biomedical Prevention
Brief Title: Pre-exposure Prophylaxis Implementation in Central-Eastern European Countries
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Columbia University (Other)
Collaborators: Yale University (Other); Fogarty International Center of the National Institute of Health (NIH)
Responsible Party: Principal Investigator, Corina Lelutiu-Weinberger, Associate Professor of Health Sciences Research (in Nursing), Columbia University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: AAAU1673; 5R33TW011752 (NIH)
Record Dates: First submitted 2022-03-25; First posted 2022-04-12 (Actual); Results first posted 2025-10-27 (Actual); Last update posted 2025-10-27 (Actual); Status verified 2025-10

CONDITIONS: Human Immunodeficiency Virus
Keywords: pre-exposure prophylaxis; gay and bisexual men
MeSH Terms: conditions — Acquired Immunodeficiency Syndrome; Homosexuality

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- PrEP Romania (Experimental): Participants will receive PrEP (as part of their standard of care), motivational counseling, and PrEP adherence support.
  Interventions: Behavioral: SPARK; Behavioral: HealthMpowerment
- Control (Active Comparator): Participants will receive PrEP (as part of their standard of care) and PrEP education during medical visits.
  Interventions: Behavioral: PrEP Education

INTERVENTIONS:
Behavioral: SPARK — SPARK is delivered in a clinic setting by a counselor using motivational interviewing techniques (e.g., open-ended questions, affirmations).
  Other Names: Sexual Health Counseling
  Arms: PrEP Romania
Behavioral: HealthMpowerment — PrEP adherence support app that utilizes engaging social networking and game-based elements, with an in-app portal for individualized live adherence counseling.
  Arms: PrEP Romania
Behavioral: PrEP Education — Educational information about PrEP provided by physician during medical visits.
  Arms: Control

SUMMARY:
To stem increasing rates of HIV among gay and bisexual men in Central-Eastern Europe, the feasibility, acceptability, and early efficacy of a culturally adapted evidence-based program to introduce pre-exposure prophylaxis (PrEP) into Romania's healthcare practice will be established. PrEP Romania, a hybrid in-person + mHealth PrEP uptake and adherence program, aims to empower gay and bisexual men and their healthcare system to adopt PrEP and support adherence. Findings can inform evidence-based PrEP rollout in other Central-Eastern European countries with similar levels of unpreparedness for biomedical prevention.

DETAILED DESCRIPTION:
Despite the effectiveness of pre-exposure prophylaxis (PrEP) in preventing HIV acquisition, PrEP is not currently medically prescribed in Romania, although demand is rapidly growing. Evidence-based knowledge is urgently needed to guide PrEP's effective rollout in Romania. First, Romania has the 2nd highest increasing HIV incidence of 15 Central-Eastern European (CEE) countries, with gay and bisexual men (GBM) being one of the few epidemic-driving groups; however, there is no national HIV programming for GBM. Second, in a large 2019 GBM report, Romania was the 8th of 44 European countries with the largest gap between PrEP use (1%) and demand (70%). Third, Romania displays some of the highest homophobic attitudes in CEE, keeping GBM in hiding and underutilizing healthcare. Consequently, many Romanian GBM obtain PrEP on their own and use it without medical guidance, thereby increasing their HIV and other health risks.

To address the unmet HIV-prevention needs of Romanian GBM, an established US-Romanian team proposes to introduce a culturally-responsive pre-exposure prophylaxis (PrEP) program in Romania. Two US-based tools will be integrated and adapted 1) SPARK, an in-person motivational intervention for uptake of and adherence to PrEP using an empowering sexual health approach; and 2) P3 (Prepared, Protected, emPowered), a PrEP adherence support app that utilizes engaging social networking and game-based elements, with an in-app portal for individualized live adherence counseling. PrEP Romania will be created with the support of a local Partner Consortium of GBM-competent health providers and community members, and be composed of both in-person (adapted SPARK to build initial motivation for PrEP uptake and adherence) and mHealth (adapted P3 to provide ongoing app-based PrEP motivation, education, and adherence support) components.

Aim 1 (R21). In months 2-11, using the ADAPT-ITT Model, SPARK and P3 will be systematically combined and culturally adapted.

Aim 2 (R21). In months 12-20, 20 GBM will be enrolled in a one-arm pilot to test PrEP Romania's feasibility (e.g., medical visit attendance), acceptability (e.g., intervention staff protocol feedback, GBM interviews about counseling, app usability, and PrEP use), and PrEP uptake (e.g., filled prescriptions), adherence (i.e., self-reported, biomarker verified) and persistence (i.e., still on PrEP) at 3 months. R21-R33 Transition Aim. In mos 21-24, PrEP Romania's promise and anticipated R33 plans will be summarized.

Aim 3 (R33). In months 1-4, necessary adjustments will be made to PrEP Romania. In months 5-30, 120 PrEP-eligible GBM in two cities will be randomized to receive either 1) PrEP Romania or 2) a PrEP education condition. Differences in PrEP adherence (self-reported and biomarker verified) between arms will be examined at 3- and 6-months post-PrEP initiation.

Aim 4 (R33). In months 31-36, individual and institutional barriers and facilitators of implementing PrEP Romania will be identified by examining Aim 3 feasibility and acceptability data, and via provider, clinic director, and GBM interviews to inform a future hybrid effectiveness-implementation trial.

ELIGIBILITY:
Men will be eligible based on CDC criteria for GBM PrEP candidates, as European guidelines are yet to be formalized:

* male sex at birth and current male identity;
* age ≥ 18;
* ≥1 acts of condomless anal sex with an HIV-positive or status-unknown male partner or diagnosis of bacterial sexually transmitted infection in past 6 months;
* intentions to start a PrEP regimen;
* confirmed to be HIV-negative upon study testing; and
* own a mobile device (smartphone, tablet, laptop); this is highly feasible given the high prevalence of smartphone and internet use in Romania, but we will cover phone plans if needed.

Exclusion Criteria:

• those not meeting eligibility

Min Age: 18 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 120 (Actual)
Dates: Start 2021-10-01 (Actual); Primary Completion 2024-09-30 (Actual); Study Completion 2024-11-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Corina Lelutiu-Weinberger, PhD, Principal Investigator — Columbia University
Locations (3):
- Columbia University School of Nursing, New York, New York, United States
- Romania (2):
  - Romanian Association Against AIDS, Bucharest
  - Romanian Association Against AIDS, Cluj-Napoca

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Lelutiu-Weinberger C, Filimon ML, Zavodszky AM, Lixandru M, Hanu L, Fierbinteanu C, Patrascu R, Streinu-Cercel A, Luculescu S, Bora M, Filipescu I, Jianu C, Hightow-Weidman LB, Rochelle A, Yi B, Buckner N, Golub SA, van Dyk IS, Burger J, Li F, Pachankis JE. Prepare Romania: study protocol for a randomized controlled trial of an intervention to promote pre-exposure prophylaxis adherence and persistence among gay, bisexual, and other men who have sex with men. Trials. 2024 Jul 10;25(1):470. doi: 10.1186/s13063-024-08313-4. PMID 38987812

RESULTS

PARTICIPANT FLOW:
Groups:
- PrEP Romania: Participants will receive PrEP, motivational counseling, and adherence support
  Pre-Exposure Prophylaxis (PrEP): FDA-approved oral medication to reduce the risk of HIV infection
  SPARK: SPARK is delivered in a clinic setting by a counselor using motivational interviewing techniques (e.g., open-ended questions, affirmations).
  HealthMpowerment: PrEP adherence support app that utilizes engaging social networking and game-based elements, with an in-app portal for individualized live adherence counseling.
- Control: Participants will receive PrEP during a medical visit.
  Pre-Exposure Prophylaxis (PrEP): FDA-approved oral medication to reduce the risk of HIV infection
  SPARK: SPARK is delivered in a clinic setting by a counselor using motivational interviewing techniques (e.g., open-ended questions, affirmations).
Period: Overall Study
Arm/Group | PrEP Romania | Control
Started | 63 | 57
Completed | 56 | 54
Not Completed | 7 | 3
Not completed — Withdrawal by Subject | 2 | 1
Not completed — Lost to Follow-up | 4 | 2
Not completed — Removed by research staff due to no longer fulfilling eligibility requirements | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | PrEP Romania | Control | Total
Number analyzed (Participants) | 63 | 57 | 120
Age, Continuous [Mean (Standard Deviation); unit: years] | 29.71 (9.44) | 28.33 (8.71) | 29.06 (9.09)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0
  Male | 63 | 57 | 120
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Romanian | 56 | 51 | 107
  Hungarian | 5 | 3 | 8
  Roma | 1 | 1 | 2
  Other | 1 | 2 | 3
Region of Enrollment [Number; unit: participants]
  Romania | 63 | 57 | 120
Study Site [Count of Participants; unit: Participants]
  Bucharest | 32 | 28 | 60
  Cluj-Napoca | 31 | 29 | 60

OUTCOME MEASURES:

1. Primary Outcome: PrEP Adherence Via Biological Measures (Binary)
Description: A binary measure of blood plasma concentration of tenofovir diphosphate (TFVdp) from PrEP medication determined using via dried blood spot or DBS analysis. ≥4 doses per week, equivalent to ≥1,000 fmol TFVdp has been shown to be protective against HIV transmission. A measurement of ≥1,000 fmol TFVdp therefore demonstrates sufficient PrEP adherence (i.e., a better outcome).
Time Frame: Measured at 3 months post-baseline and 6 months post-baseline
Population: Some participants were lost to follow-up, and in some cases participants did not provide data for certain outcomes on self-administered surveys or via blood testing. Therefore, at some timepoints, "Number Analyzed" may be less that 63 for PrEP Romania arm and 57 for Control arm.
Measure: Count of Participants; unit: Participants
Arm/Group | PrEP Romania | Control
Number analyzed (Participants) | 63 | 57
Participants
  3 months post-baseline: number analyzed (Participants) | 58 | 53
  3 months post-baseline: >= 1000 fmol TFVdp | 47 | 34
  3 months post-baseline: < 1000 fmol TFVdp | 11 | 19
  6 months post-baseline: number analyzed (Participants) | 52 | 52
  6 months post-baseline: >= 1000 fmol TFVdp | 38 | 30
  6 months post-baseline: < 1000 fmol TFVdp | 14 | 22

2. Secondary Outcome: PrEP Adherence Via Biological Measures (Continuous)
Description: A continuous measure of blood plasma concentration of tenofovir diphosphate (TFVdp) from PrEP medication determined using via dried blood spot (DBS) analysis. A higher measure of fmol TFVdp demonstrates greater PrEP adherence (i.e., a better outcome).
Time Frame: Measured at 3 months post-baseline and 6 months post-baseline
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: fmol TFVdp
Arm/Group | PrEP Romania | Control
Number analyzed (Participants) | 63 | 57
fmol TFVdp
  3 months post-baseline: number analyzed (Participants) | 58 | 53
  3 months post-baseline | 1963.98 (1194.07) | 1867.45 (1452.07)
  6 months post-baseline: number analyzed (Participants) | 52 | 52
  6 months post-baseline | 1777.38 (1162.16) | 1481.46 (1373.62)

3. Secondary Outcome: PrEP Adherence Via Self-report Measures (Binary)
Description: A binary measure of PrEP adherence obtained from participant self-report data. Each week, participants mark the days over the past week on which they took or missed their PrEP dose. Each participant's weekly survey results are averaged to determine their mean number of PrEP doses taken per week over the past 3 months. The binary version of this outcome is defined as: 0-3 doses per week, on average, vs. ≥4 doses per week, on average, with ≥4 doses representing a sufficient level of PrEP adherence to be protected against HIV transmission (i.e., a better outcome).
Time Frame: Measured at 3 months post-baseline and 6 months post-baseline.
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | PrEP Romania | Control
Number analyzed (Participants) | 63 | 57
Participants
  3 months post-baseline: number analyzed (Participants) | 57 | 54
  3 months post-baseline: >=4 doses per week, on average | 56 | 54
  3 months post-baseline: 0-3 doses per week, on average | 1 | 0
  6 months post-baseline: number analyzed (Participants) | 54 | 54
  6 months post-baseline: >=4 doses per week, on average | 53 | 52
  6 months post-baseline: 0-3 doses per week, on average | 1 | 2

4. Secondary Outcome: PrEP Adherence Via Self-report Measures (Continuous)
Description: A continuous measure of PrEP adherence obtained from participant self-report data. Each week, participants mark the days over the past week on which they took or missed their PrEP dose. Each participant's weekly survey results are averaged to determine their mean number of PrEP doses taken per week over the past 3 months, with higher numbers indicating greater PrEP adherence (i.e., a better outcome).
Time Frame: Measured at 3 months post-baseline and 6 months post-baseline.
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: doses per week
Arm/Group | PrEP Romania | Control
Number analyzed (Participants) | 63 | 57
doses per week
  3 months post-baseline: number analyzed (Participants) | 57 | 54
  3 months post-baseline | 6.72 (0.86) | 6.81 (0.49)
  6 months post-baseline: number analyzed (Participants) | 54 | 54
  6 months post-baseline | 6.62 (0.99) | 6.43 (1.00)

5. Secondary Outcome: PrEP Motivation
Description: PrEP motivation is assessed through participants responses to a single question ("If you are using/were to use PrEP, how motivated are you/would you be to take the pill every day?") with responses scored from 1 to 7 (1=not at all motivated 7=extremely motivated). Higher scores indicate greater PrEP motivation (i.e., a better outcome).
Time Frame: Measured at baseline, 3 months post-baseline, and 6 months post-baseline
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | PrEP Romania | Control
Number analyzed (Participants) | 63 | 57
score on a scale
  Baseline | 6.52 (1.22) | 6.47 (0.93)
  3 months post-baseline: number analyzed (Participants) | 62 | 56
  3 months post-baseline | 6.29 (1.53) | 6.07 (1.33)
  6 months post-baseline: number analyzed (Participants) | 58 | 55
  6 months post-baseline | 6.48 (0.94) | 6.09 (1.22)

6. Secondary Outcome: PrEP Knowledge
Description: PrEP knowledge is measured through 3 multiple choice questions about PrEP efficacy (e.g., "If taken as indicated by the provider, how effective is PrEP at preventing HIV infection?") where responses are scored as 0 (incorrect or unsure) or 1 (correct). Participants responding correctly to all 3 questions are assigned a total score of 1 (higher PrEP knowledge (i.e., a better outcome)), whereas all others are assigned a total score of 0.
Time Frame: Measured at baseline, 3 months post-baseline, and 6 months post-baseline
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | PrEP Romania | Control
Number analyzed (Participants) | 63 | 57
Participants
  Baseline: 1 (all correct) | 40 | 27
  Baseline: 0 (not all correct) | 23 | 30
  3 months post-baseline: number analyzed (Participants) | 62 | 56
  3 months post-baseline: 1 (all correct) | 42 | 37
  3 months post-baseline: 0 (not all correct) | 20 | 19
  6 months post-baseline: number analyzed (Participants) | 58 | 55
  6 months post-baseline: 1 (all correct) | 35 | 37
  6 months post-baseline: 0 (not all correct) | 23 | 18

7. Secondary Outcome: PrEP Attitudes and Beliefs - Positive Statements Subscore
Description: Pro-PrEP attitudes and beliefs are measured via a 3-item scale scale consisting of statements describing favorable opinions about PrEP (e.g., "A daily pill would be a good way to protect myself against HIV"). Respondents mark their level of agreement with each item on a scale from 1 (totally disagree) to 5 (totally agree). The 3 individual item scores are summed to obtain an overall score from 5-15, where higher overall scores indicate greater positive attitudes/beliefs about PrEP (i.e., a better outcome).
Time Frame: Measured at baseline, 3 months post-baseline, and 6 months post-baseline
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | PrEP Romania | Control
Number analyzed (Participants) | 63 | 57
score on a scale
  Baseline | 14.57 (1.20) | 14.56 (0.95)
  3 months post-baseline: number analyzed (Participants) | 62 | 56
  3 months post-baseline | 14.60 (0.86) | 14.34 (1.21)
  6 months post-baseline: number analyzed (Participants) | 58 | 53
  6 months post-baseline | 14.55 (0.98) | 14.49 (1.05)

8. Secondary Outcome: PrEP Attitudes and Beliefs - Negative Statements Subscore
Description: Negative PrEP attitudes and beliefs are measured via a 7-item scale scale consisting of statements describing negative opinions about PrEP (e.g., " I would be very embarrassed to take HIV medication if I didn't have HIV"). Respondents mark their level of agreement with each item on a scale from 1 (totally disagree) to 5 (totally agree). The 7 individual item scores are summed to obtain an overall score from 7-35, where higher overall scores indicate greater negative attitudes/beliefs about PrEP (i.e., a worse outcome).
Time Frame: Measured at baseline, 3 months post-baseline, and 6 months post-baseline
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | PrEP Romania | Control
Number analyzed (Participants) | 63 | 57
score on a scale
  Baseline | 14.76 (3.29) | 14.19 (4.65)
  3 months post-baseline: number analyzed (Participants) | 62 | 55
  3 months post-baseline | 14.13 (3.06) | 14.49 (4.63)
  6 months post-baseline: number analyzed (Participants) | 57 | 52
  6 months post-baseline | 13.95 (3.77) | 14.27 (4.49)

9. Secondary Outcome: PrEP Barriers
Description: Barriers to taking PrEP are measured via an 11-item scale scale consisting of statements describing potential barriers to taking PrEP (e.g., "the fact that you have to take a pill every day"). Respondents mark the degree to which each item is important to them on a scale from 1 (not important at all) to 5 (extremely important). The 11 individual item scores are summed to obtain an overall score from 11-55, where higher overall scores indicate more barriers to taking PrEP (i.e., a worse outcome).
Time Frame: Measured at baseline, 3 months post-baseline, and 6 months post-baseline
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | PrEP Romania | Control
Number analyzed (Participants) | 63 | 57
score on a scale
  Baseline | 23.05 (8.47) | 25.67 (8.49)
  3 months post-baseline: number analyzed (Participants) | 62 | 56
  3 months post-baseline | 21.92 (8.05) | 25.21 (8.40)
  6 months post-baseline: number analyzed (Participants) | 58 | 53
  6 months post-baseline | 22.67 (7.92) | 23.94 (7.96)

10. Secondary Outcome: PrEP Facilitators
Description: Facilitators for taking PrEP are measured via an 8-item scale scale consisting of statements describing potential facilitators for taking PrEP (e.g., "the fact that I don't have to pay for PrEP"). Respondents mark the degree to which each item is important to them on a scale from 1 (not important at all) to 5 (extremely important). The 8 individual item scores are summed to obtain an overall score from 8-40, where higher overall scores indicate more facilitators for taking PrEP (i.e., a better outcome).
Time Frame: Measured at baseline, 3 months post-baseline, and 6 months post-baseline
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | PrEP Romania | Control
Number analyzed (Participants) | 63 | 57
score on a scale
  Baseline | 33.14 (6.64) | 35.12 (4.31)
  3 months post-baseline: number analyzed (Participants) | 62 | 56
  3 months post-baseline | 34.31 (5.14) | 35.27 (5.05)
  6 months post-baseline: number analyzed (Participants) | 58 | 53
  6 months post-baseline | 34.66 (5.38) | 35.38 (4.64)

11. Secondary Outcome: PrEP Stigma - Score on PrEP Stigma Scale-Shortened Version
Description: The PrEP Stigma Scale-Shortened Version is an 11 item scale measuring anticipated and/or perceived stigma related to PrEP use. Participants state their level of agreement (1=strongly disagree, 5=strongly agree) to statements about PrEP-related stigma (e.g., "My friends would think less of me if they found out I was using PrEP"). Item scores are summed to obtain an overall score from 11 to 55, with higher total scores indicate increased stigma (i.e., a worse outcome).
Time Frame: Measured at baseline, 3 months post-baseline, and 6 months post-baseline
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | PrEP Romania | Control
Number analyzed (Participants) | 63 | 57
score on a scale
  Baseline | 19.68 (5.95) | 20.19 (8.53)
  3 months post-baseline: number analyzed (Participants) | 62 | 56
  3 months post-baseline | 18.63 (6.50) | 19.91 (8.11)
  6 months post-baseline: number analyzed (Participants) | 58 | 53
  6 months post-baseline | 18.59 (7.57) | 19.15 (7.91)

12. Secondary Outcome: Depression Symptomology - Score on Patient Health Questionnaire-9 Item (PHQ-9)
Description: The Patient Health Questionnaire-9 item (PHQ-9) measures severity of depression symptoms in the last 2 weeks, with respondents quantifying the frequency (0=not at all, 3=nearly every day) of their depression symptoms (e.g., Little interest or pleasure in doing things). Item scores are summed to obtain an overall score from 0-27 with higher overall scores indicate increased depression symptoms (i.e., a worse outcome).
Time Frame: Measured at baseline, 3 months post-baseline, and 6 months post-baseline
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | PrEP Romania | Control
Number analyzed (Participants) | 63 | 57
score on a scale
  Baseline | 4.35 (5.38) | 5.42 (5.55)
  3 months post-baseline: number analyzed (Participants) | 62 | 56
  3 months post-baseline | 3.55 (4.03) | 3.29 (3.70)
  6 months post-baseline: number analyzed (Participants) | 58 | 53
  6 months post-baseline | 4.69 (6.19) | 4.55 (5.04)

13. Secondary Outcome: Anxiety Symptomology - Score on Generalized Anxiety Disorder 7-item(GAD-7)
Description: The Generalized Anxiety Disorder 7-item(GAD-7) measures severity of anxiety symptoms in the last 2 weeks, with respondents quantifying the frequency (0=not at all, 3=nearly every day) of their anxiety symptoms (e.g., Feeling nervous, anxious or on edge). Item scores are summed to obtain an overall score from 0-21 with higher overall scores indicate increased anxiety symptoms (i.e., a worse outcome).
Time Frame: Measured at baseline, 3 months post-baseline, and 6 months post-baseline
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | PrEP Romania | Control
Number analyzed (Participants) | 63 | 57
score on a scale
  Baseline | 3.86 (4.35) | 4.33 (4.86)
  3 months post-baseline: number analyzed (Participants) | 62 | 56
  3 months post-baseline | 2.69 (3.48) | 2.36 (2.71)
  6 months post-baseline: number analyzed (Participants) | 58 | 53
  6 months post-baseline | 3.48 (4.62) | 3.34 (3.88)

14. Secondary Outcome: HIV Risk - Number of Condomless Anal Sex (CAS) Acts
Description: HIV risk, measured by number of condomless anal sex (CAS) acts with an HIV-positive or status-unknown male partner over the past 6 months is self-reported by participants. A higher number of CAS acts represents greater HIV risk (i.e., a worse outcome).
Time Frame: Baseline and 6 months post-baseline
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: condomless anal sex acts
Arm/Group | PrEP Romania | Control
Number analyzed (Participants) | 63 | 57
condomless anal sex acts
  Baseline | 23.60 (34.25) | 21.00 (23.10)
  6 months post-baseline: number analyzed (Participants) | 58 | 53
  6 months post-baseline | 18.21 (28.72) | 10.04 (15.45)

15. Secondary Outcome: Sexually Transmitted Infection (STI) Diagnoses
Description: Participants were asked whether they had been diagnosed with any bacterial sexually transmitted infections (STIs) over the past 6 months. This self-reported measure was coded in a binary manner as either yes (i.e., a worse outcome) or no.
Time Frame: Baseline and 6 months post-baseline
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | PrEP Romania | Control
Number analyzed (Participants) | 63 | 57
Participants
  Baseline: Yes | 24 | 18
  Baseline: No | 39 | 39
  6 months post-baseline: number analyzed (Participants) | 58 | 53
  6 months post-baseline: Yes | 13 | 15
  6 months post-baseline: No | 45 | 38

ADVERSE EVENTS:
Time Frame: During an assessment, from baseline survey to 6 months post-baseline
Description: Participants were assessed as soon as a trigger was sent to the team by a score in a survey.
Arm/Group | PrEP Romania | Control
All-Cause Mortality (participants affected / at risk) | 0/63 | 0/57
Serious Adverse Events (participants affected / at risk) | 1/63 | 0/57
Other Adverse Events (participants affected / at risk) | 6/63 | 8/57
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | PrEP Romania (N=63) | Control (N=57)
Hospitalization (Infections and infestations) | 1 (1) | 0 (0) — Participant hospitalized overnight for infection whose cause was unrelated to study participation.
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | PrEP Romania (N=63) | Control (N=57)
Suicidal ideation (Psychiatric disorders) | 6 (6) | 8 (8)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2024-07-10): https://cdn.clinicaltrials.gov/large-docs/23/NCT05323123/Prot_000.pdf
  • Statistical Analysis Plan (2025-09-18): https://cdn.clinicaltrials.gov/large-docs/23/NCT05323123/SAP_001.pdf